CLINICAL TRIAL: NCT07293637
Title: Identifying the Neural Correlates of Mental Simulation in Multi-Step Planning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24-1331; 1R01MH134979-01A1 (NIH)
Record Dates: First submitted 2025-12-17; First posted 2025-12-19 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Decision Making; Cognition; Mental Simulation; Problem Solving; Planning
Keywords: Four-in-a-Row; Planning; Tree search; Computational modeling; Eye tracking; MEG; fMRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MEG cohort (Experimental): Single-group study in healthy adults. Participants complete a behavioral training session and then an in-person session performing the Four-in-a-Row planning task during MEG (with an additional MEG localizer task, as applicable).
  Interventions: Behavioral: Four-in-a-Row Task

INTERVENTIONS:
Behavioral: Four-in-a-Row Task — Deterministic, adversarial 'Four-in-a-Row' decision-making task that requires thinking multiple steps ahead. Participants complete a training/gameplay session and a laboratory session in which they choose moves from mid-game positions while behavioral responses (and eye movements, if applicable) are recorded. After the neuroimaging session, participants may play a full match outside the scanner for an additional monetary reward.

SUMMARY:
Planning is the ability to think ahead by considering possible future actions and their consequences. This research study aims to understand how the brain supports multi-step planning by testing whether people simulate promising future move sequences while deciding what to do next. Healthy adult volunteers will learn and play a strategy game called "Four-in-a-Row" (similar to Connect Four). Participants will complete two sessions on successive days: an online behavioral training/playing session and an in-person brain-recording session at New York University. During the brain-recording session, participants will view mid-game board positions and choose the best move while the study team records brain activity (using magnetoencephalography [MEG] or functional MRI [fMRI]) and eye movements. Data from the game and eye tracking will also be used to fit computational models of planning that help interpret the neural measurements.

DETAILED DESCRIPTION:
This is a human neuroimaging study consisting of two related experiments designed to characterize the neural correlates of mental simulation during multi-step planning in the "Four-in-a-Row" game. Planning is modeled as a feature-based heuristic evaluation combined with look-ahead (tree search) that evaluates candidate actions by simulating future states and outcomes.

Participants complete two sessions on successive days. Session 1 is a ~60-minute online behavioral session in which participants learn the rules of Four-in-a-Row (including a comprehension/quiz check) and play multiple games against computer opponents spanning difficulty levels. Behavioral data from Session 1 are used to fit a computational model of planning for each participant.

Session 2 is an in-person neuroimaging session with simultaneous eye tracking. In the MEG experiment, participants complete a feature localizer followed by a primary planning task in which they evaluate mid-game board positions with a fixed decision window (e.g., 15 seconds) to encourage planning. B2 In the fMRI experiment, participants complete a planning task while BOLD activity and eye movements are recorded, using a trial structure designed to dissociate model-derived quantities such as myopic value and tree-search value.

The main analyses will test where (fMRI) and when (MEG) the brain represents simulated future states, their values, and the evolving decision process, guided by participant-specific computational-model predictions.

ELIGIBILITY:
Inclusion Criteria:

* N/A

Exclusion Criteria:

* History of neurological or psychiatric illness
* Vulnerable populations

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percent of moves correctly predicted by the behavioral model | 1 hour
  Participant choices in the Four-in-a-Row task are used to fit a computational behavioral model. After fitting, the model predicts an action for each state; we quantify the percent of participant moves matched by the model's predicted move.
MEG activity | 1 hour
  Task-evoked MEG activity during different stages of the task, specifically deliberation about upcoming decisions.

CONTACTS AND LOCATIONS:
Locations (1):
- New York University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level behavioral task data (choices/RT), eye-tracking measures, and analysis code. Neuroimaging data will be shared as de-identified derivatives (and/or raw data if allowed by consent and de-identification procedures). Supporting metadata/documentation (e.g., scanning protocols) and analytic code used for published analyses will also be shared.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: IPD and supporting information will be made available starting 12 months after the NIH award begins, with updates deposited every 6 months thereafter, and will remain available indefinitely.
Access Criteria: De-identified IPD will be available through the NIMH Data Archive (NDA) and via OSF/OpenNeuro for relevant datasets, with analytic code shared via GitHub. We will not impose any investigator-specific limitations on access, distribution, or reuse beyond standard repository requirements (e.g., account registration and agreement to repository terms). All shared data will be de-identified.
URL: https://nda.nih.gov

DOCUMENTS (1):
  • Informed Consent Form (2025-12-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT07293637/ICF_000.pdf